CLINICAL TRIAL: NCT06368648
Title: An Early Feasibility Study for the Development of a Model to Non-Invasively Estimate Intracranial Pressure (ICP) and New Metrics of Cerebral Autoregulation (CAR) Using the CoMind One EFS Device
Brief Title: CoMind Early Feasibility Study
Acronym: CoMind EFS
Status: Recruiting | Type: Observational
Sponsor: CoMind Technologies Limited (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Intracranial Pressure; Intracranial Pressure Changes; Traumatic Brain Injury; Intracerebral Hemorrhage; Encephalitis; Encephalopathy; Hydrocephalus; Stroke; Autoregulation
Keywords: Intracranial Pressure; Traumatic Brain Injury; Cerebral Autoregulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage; Encephalitis; Brain Diseases; Hydrocephalus; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving invasive ICP and ABP monitoring as their standard of care: Patients who are receiving invasive Intracranial Pressure (ICP) monitoring and invasive Arterial Blood Pressure (ABP) monitoring as per standard practice will serve as their own controls.

SUMMARY:
The purpose of this research, which has been determined as non-significant risk by the central IRB overseeing the study, is to obtain information to help further develop a machine (a medical device) to measure the pressure around the brain from the outside (this pressure is called intracranial pressure or ICP). Monitoring and managing ICP is an important part of care for patients with conditions such as Traumatic Brain Injury (TBI). However, the current way of measuring ICP requires surgery to drill a hole into the skull, and therefore can introduce additional risks such as infections and pain.

Recent research has shown it may be possible to measure ICP without needing surgery. This technology is in development, but large amounts of data is required to build these new devices.

Through collecting a large database of information from patients who have both the routine surgical device and the research device applied to their head, the research team will work to develop and test an effective and potentially safer way of monitoring patient ICP.

DETAILED DESCRIPTION:
A prospective, observational study, determined as non-significant risk by the Central IRB, to assess and improve performance of a non-invasive ICP estimation system. The development of non-invasive systems is intended to replace the need for invasive ICP monitors. Participants serve as their own controls with concurrent, synchronous measurements of ICP (measured invasively as per standard clinical practice), Arterial Blood Pressure (ABP- measured invasively as per standard clinical practice), and measurements of a novel non- invasive cerebral blood-flow index (CBFi) from the CoMind One EFS device. These signals will be recorded simultaneously. The ABP and CBFi will serve as inputs to a model which outputs a non-invasive estimate of ICP, and the invasive ICP signal will be used to supervise and evaluate the performance of the non-invasive ICP estimation model. A large volume of data shall be collected for the purposes of training and testing the non-invasive ICP model. The Sponsor will report limits of agreement (LOA) between data-driven estimates of ICP and the invasively measured signal. In addition, this study will compare metrics built on non-invasive estimation of ICP or CBFi that indicate the state of CAR, and the limits of Autoregulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female sex at birth, and aged 18 years or older on the date of enrollment.
2. Receiving continuous invasive ICP monitoring (Bolt or EVD) as part of standard care.
3. Invasive ICP monitor catheter penetrating the parenchyma or ventricles.
4. Receiving continuous invasive ABP monitoring as part of standard care.

Exclusion Criteria:

1. Presence of any implant (cosmetic or otherwise) in the frontal bone in such proximity to the CoMind One EFS Sensor that they might physically touch.
2. Open wounds on the forehead such that CoMind One EFS Sensor cannot be safely placed over an area of intact skin
3. Presenting with radiographic evidence of a non-intact skull at the recording site on admission.
4. If patient is enrolled in an intervention/study that may interfere with SoC ICP measurements or the CoMind One EFS device measurement then the patient is ineligible.
5. Patients with decompressive craniectomy will be excluded unless a CoMind One EFS recording can be made from intact skull.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any participant (18 years or older) who is undergoing invasive ICP monitoring and continuous ABP monitoring as part of their normal medical treatment at selected clinical sites. The majority of such participants will have sustained a Traumatic Brain Injury (TBI), but some may have Intracerebral Haemorrhage (ICH), Encephalitis, various metabolic Encephalopathies (notably hepatic), Hydrocephalus (both communicating and non-communicating), or Stroke, although this is not an exhaustive list of participant conditions.
Sampling Method: Non-Probability Sample
Enrollment: 581 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
A test of the difference in estimation errors between two non-invasive ICP estimation models: one trained with ABP and CoMind One EFS CBFi, and one trained only using ABP | From enrollment to the end of observation (either 3 weeks after removal of the CoMind device or until ICU discharge, whichever event is sooner)
Models trained using CoMind CBFi and ABP will be evaluated based on their limits of agreement (LOA) with invasive ICP. | From enrollment to the end of observation (either 3 weeks after removal of the CoMind device or until ICU discharge, whichever event is sooner)
  The threshold limit of agreement will be evaluated at three levels corresponding to a model with clinical utility that is optimal, high, or moderate clinical utility. These levels of clinical utility are defined as follows: ● Optimal clinical utility: a model trained using CoMind CBFi and ABP can achieve LOA with invasive ICP less-than or equal to +/-2 mmHg in the range of ICP between 10-30 mmHg, and less-than or equal to +/-4 mmHg in the ranges of 0-10 mmHg, and 30-50 mmHg. ● High clinical utility: a model trained using CoMind CBFi and ABP can achieve LOA with invasive ICP less-than or equal to +/-3 mmHg in the range of ICP between 10-30 mmHg, and less-than or equal to +/-5 mmHg in the ranges of 0-10 mmHg, and 30-50 mmHg. ● Moderate clinical utility: a model that achieves LOA with invasive ICP less-than or equal to +/-4 mmHg in the range of ICP between 10-30 mmHg, and less-than or equal to +/-6 mmHg in the ranges of 0-10 mmHg, and 30-50 mmHg.

SECONDARY OUTCOMES:
Demonstration that non-invasive ICP estimation using the CoMind One EFS device is insensitive to differences in skin tone across the population. | From enrollment to the end of observation (either 3 weeks after removal of the CoMind device or until ICU discharge, whichever event is sooner)
Demonstration of a non-invasive ICP model that can classify the transition between ICP 'states', i.e. transitions between low ICP (less than 20 mmHg), and high ICP (greater than 20 mmHg). | From enrollment to the end of observation (either 3 weeks after removal of the CoMind device or until ICU discharge, whichever event is sooner)
Demonstration of a non-invasive ICP waveform prediction model and assessment of its accuracy against the invasively-measured ICP waveform. | From enrollment to the end of observation (either 3 weeks after removal of the CoMind device or until ICU discharge, whichever event is sooner)
Demonstration of an non-invasive ICP model that can predict trends in ICP | From enrollment to the end of observation (either 3 weeks after removal of the CoMind device or until ICU discharge, whichever event is sooner)

OTHER OUTCOMES:
A comparison of metrics of CAR derived from CoMind One EFS CBFi, CoMind One EFS device estimates of ICP, and ABP. | From enrollment to the end of observation (either 3 weeks after removal of the CoMind device or until ICU discharge, whichever event is sooner)

CONTACTS AND LOCATIONS:
Overall Officials: Ramani Balu, MD, PhD, Principal Investigator — Inova Fairfax Hospital
Locations (11):
- United States (11):
  - UC Davis Medical Center, Sacramento, California
  - Christiana Care, Wilmington, Delaware
  - Jackson Memorial Hospital, Miami, Florida
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Washington University Medical Center, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - WakeMed, Raleigh, North Carolina
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - University of Washington, Harborview, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No